CLINICAL TRIAL: NCT07079540
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Active-Controlled Parallel Group Phase III Clinical Study to Evaluate the Efficacy and Safety of X842 Capsules in Patients With Reflux Esophagitis
Brief Title: The Phase III Clinical Trial of X842 Capsules for Reflux Esophagitis
Acronym: X842
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Sinorda Biomedicine Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SND-X842-301; ChiCTR20210736 (Other: ChiCTR)
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Reflux Esophagitis
Keywords: Reflux Esophagitis; X842; Population Pharmacokinetics, PopPK; Lansoprazole
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Lansoprazole

STUDY DESIGN:
Intervention Model Description: After completing the relevant laboratory tests and endoscopic examinations at screening, subjects who meet the inclusion criteria and do not meet the exclusion criteria are randomly under blinding at a 3:1 ratio assigned to test group(X842 Capsule)and control group ( Lansoprazole enteric-coated Capsules) for for 4-week treatment and then receive endoscopy. If endoscopy shows healed esophagitis, treatment will be discontinued; if esophagitis remains unhealed, treatment continues for an additional 4 weeks. The minimum treatment duration with either test or control drug is 4 weeks, and the maximum is 8 weeks in this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial uses a double-blind double-dummy design, where the investigator, the subject and the other parties involved in the trial are blinded to the drug given to the subject. X842 capsules (test group)and and placebo, lansoprazole enteric-coated capsules (control group)and placebo, are provided by Jiangsu Sinorda Biomedicine Co., Ltd. The physical appearance, shape, specification and dosage of the test drug and comparator as well as the placebo are generally similar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- X842 50mg QD (Experimental): X842 50 mg, capsule, orally, once daily and lansoprazole placebo-matching capsule, orally, once daily up to 4 to 8 weeks.
  Interventions: Drug: X842; Drug: Lansoprazole Placebo
- lansoprazole 30mg QD (Active Comparator): Lansoprazole 30 mg, capsule, orally, once daily and X842 placebo-matching capsule, orally, once daily up to 4 weeks.
  Interventions: Drug: X842 Placebo; Drug: Lansoprazole

INTERVENTIONS:
Drug: X842 — X842 capsules
  Other Names: X842 capsules
  Arms: X842 50mg QD
Drug: X842 Placebo — X842 placebo-matching capsules
  Arms: lansoprazole 30mg QD
Drug: Lansoprazole — Lansoprazole capsules
  Other Names: Lansoprazole capsules
  Arms: lansoprazole 30mg QD
Drug: Lansoprazole Placebo — Lansoprazole placebo-matching capsules
  Arms: X842 50mg QD

SUMMARY:
To evaluate the efficacy and safety of X842 Capsules 50 mg compared to Lansoprazole Enteric Capsules for the treatment of reflux esophagitis, and to characterize the population pharmacokinetics of X842 capsules in this patient population.

DETAILED DESCRIPTION:
This study uses a multicenter, randomized, double-blind, double-dummy, active-controlled parallel-group, non-inferiority design to compare the efficacy and safety of X842 capsules (50 mg) in the treatment of reflux esophagitis over 4 to 8 weeks in comparison with lansoprazole enteric-coated capsules(30 mg) . Additionally, the population pharmacokinetics characteristics of X842 capsules in patients with reflux esophagitis is observed.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 years ≤ age ≤ 75 years;
2. Within 7 days prior to randomization, the subjects are endoscopically diagnosed with reflux esophagitis from Los Angeles (LA) grade A to D (notes: the percent of the subjects with LA grade A of RE should be no more than 20% of the all subjects who are planned to be enrolled in the study);
3. Subjects who can independently complete the subject diary cards;
4. Subjects fully understand the trial contents, participate in the trial voluntarily, and sign the informed consent forms.

Exclusion Criteria:

1. Subjects who receive X842 capsules or other P-CAB drugs in previous clinical studies;
2. Subjects known to be allergic to X842 capsules or lansoprazole enteric-coated capsules, or relevant excipients of X842 capsules or lansoprazole enteric-coated capsules, such as lactose, microcrystalline cellulose, croscarmellose sodium, sodium dodecyl sulfate, sodium stearyl fumarate, and silicon dioxide;
3. Subjects unable to receive upper gastrointestinal endoscopy;
4. Endoscopic examination revealed concomitant diseases potentially affecting the esophagus, excluding hiatal hernia, and excluding Barrett's esophagus with metaplastic columnar epithelium that either does not involve the entire esophageal circumference or is short-segment (< 3 cm in length).
5. Patients with rheumatic/autoimmune diseases potentially affecting esophageal motility (e.g., scleroderma, undifferentiated connective tissue disease), or those with a history of esophageal radiotherapy or cryotherapy;
6. Subjects who have acute upper gastrointestinal hemorrhage within 4 weeks prior to enrollment;
7. Subjects with active peptic ulcer discovered during upper gastrointestinal endoscopy, or subjects with suspicious or definite malignancies;
8. Subjects known to have Zollinger-Ellison syndrome or inflammatory bowel disease (IBD);
9. Subjects with history of surgery affecting the structure or function of the esophagus, stomach, or duodenum, or surgery altering gastric acid secretion.
10. Subjects who plan to undergo surgical procedures during the study period that may alter gastric acid secretion (e.g., abdominal surgery, vagotomy, or craniectomy).
11. Subjects with a history of malignancies within 5 years prior to screening (a subject can participate in the study if his /her skin basal cell carcinoma or carcinoma in situ of uterine cervix has been cured);
12. Subjects with concomitant serious diseases of central nervous system, cardiovascular system, respiratory system, liver, kidney, gastrointestinal tract, urinary system, endocrine system, or hematological system, and the investigator thinks these diseases may mix the study results up or affect the safety of the subject;
13. Laboratory test results at screening showing that ALT or AST is larger than 1.5 times of the upper limit of normal, or kidney function index Cr is larger than the upper limit of normal (a re-examination is permitted in the study, and subjects will be excluded if they still fail to meet the inclusion criteria);
14. Subjects who use of therapeutic doses of GERD medications within 7 days prior to randomization, eg. proton pump inhibitors (PPIs), P-CABs, histamine2 receptor antagonists (H2RAs), or gastric mucosal protectors (except hydrotalcite), prokinetic drugs, and traditional Chinese medicines;
15. Subjects who chronically use non-steroidal anti-inflammatory drug (including cyclooxygenase-2 inhibitor), anti-platelet drug (such as aspirin and clopidogrel), or anticoagulant (such as Warfarin) prior to randomization, and can not stop the medication during the trial;
16. At screening, subjects with clinically significant ECG abnormalities, including serious arrhythmia, multifocal ventricular premature complexes, grade II or above atrioventricular block, and prolongation of the Q-Tc interval (QTc≥450 ms in males and QTc≥470 ms in females);
17. Subjects who are using atazanavir sulfate or ripivirin hydrochloride at screening;
18. Subjects with a history of long-term abuse of drug or alcohol within 6 months prior to screening;
19. Female subjects with known pregnancy, those in breast-feeding period, or those who are planned to become pregnant during the trial. At the investigator's discretion, women of childbearing age who cannot use a medically-proven and reliable method of contraception from signing the informed consent forms to 4 weeks after the last dose of the study;
20. Subjects who participate in other drug/medical device clinical studies and use the drug/medical device within 3 months prior to randomization;
21. Subjects who are considered unsuitable for participating in this trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects Whose Reflux Esophagitis is Cured as Confirmed by Endoscopy at Week 8 | 8 weeks
  Healing of reflux esophagitis is defined as endoscopic confirmation of resolved esophagitis (absence of esophageal mucosal breaks) in subjects.

SECONDARY OUTCOMES:
Proportion of Subjects Whose Reflux Esophagitis is Cured as Confirmed by Endoscopy at Week 4 | 4 weeks
  Healing of reflux esophagitis is defined as endoscopic confirmation of resolved esophagitis (absence of esophageal mucosal breaks) in subjects.
Improvement rate in the frequency and severity of individual clinical symptoms (heartburn, regurgitation) of reflux esophagitis at Weeks 2, 4, and 8 after treatment initiation. | 2,4,8 weeks
  Improvement in the frequency of clinical symptom occurrence: Defined as subjects whose symptom frequency score before treatment was ≥1 point had a reduction of ≥1 point after treatment compared to before treatment.
  Improvement in the severity of clinical symptoms: Defined as a reduction of ≥1 point in the symptom severity score of subjects with a score of ≥1 point before treatment after treatment compared to before treatment.
Response rates for individual symptom domains (heartburn, regurgitation) in reflux esophagitis at Weeks 2, 4, and 8 post-baseline. | 2.4.8 weeks
  Resolution of individual clinical symptoms: defined as the achievement of score 0 in both severity and frequency for symptoms with baseline scores ≥1.
Overall symptomatic resolution rate for reflux esophagitis at Weeks 2, 4, and 8 | 2,4,8 weeks
  Overall Clinical Symptom Resolution: Defined as the achievement of a score of 0 (i.e., complete disappearance) for all symptoms of reflux esophagitis in subjects with any individual symptom score ≥1 at baseline.
Change in serum gastrin levels from baseline at Weeks 4 and 8 of treatment | 4, 8 weeks
  Serum gastrin testing will be conducted at the central laboratory. The change between the serum gastrin values collected at Weeks 4 and 8 relative to baseline.
Number of Subjects Reporting Who Had One or More Treatment-emergent Adverse Event (TEAE) | up to 8 weeks
  Adverse event is defined as any adverse medical event that is observed in a subject who is receiving a drug treatment or in a clinical study, and that does not necessarily have a causal relationship with the treatment.
Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of blood serum Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of blood serum | up to 8 weeks
  Number of subjects with any markedly abnormal values in laboratory tests of blood serum collected throughout study is reported.
Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of blood | up to 8 weeks
  Number of subjects with any markedly abnormal values in laboratory tests of blood collected throughout study is reported.
Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of urine | up to 8 weeks
  Number of subjects with any markedly abnormal values in laboratory tests of urine collected throughout study is reported.collected throughout study is reported.
Number of Subjects With Markedly Abnormal Electrocardiogram (ECG) Findings | up to 8 weeks
  The investigator or the sub-investigator interpreted the ECG using one of the following categories: "within normal limits", "abnormal but not clinically significant", or "abnormal and clinically significant"
Vital signs | up to 8 weeks
  Blood pressure, respiration, heart rate and body temperature were evaluated at each visit during the screening period and the double-blind treatment period
Pharmacokinetic evaluation | up to 8 weeks
  Quantification of plasma concentrations of X842 and its metabolites to characterize the population pharmacokinetic profile of X842 capsules in GERD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Hu, Ph.D, Study Chair — Jiangsu Sinorda Biomedicine Co., Ltd
Locations (53):
- China (53):
  - Liuan People's Hospital, Liu‘an, Anhui
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - The 900th Hospital of the Joint Logistic Support Force of the People's Liberation Army of China, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The Second Nanning People's Hospital, Nanjing, Guangxi
  - The Affiliated Hospital of Guzihou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital of Shiyan City, Shiyan, Hubei
  - Affiliated Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Chenzhou City, Chenzhou, Hunan
  - The Second Affiliated Hospital of South China University, Hengyang, Hunan
  - The First Affiliated Hospital Of University Of South China, Hengyang, Hunan
  - Huai 'an First People's Hospital, Huaian, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Zhongda Hospital of Southeast University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Yangzhou University(Yangzhou First People's Hospital), Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jinlin
  - The First Hospital of Jilin University, Changchun, Jinlin
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Affiliated Hospital of Binzhou Medical University, Binzhou, Shandong
  - Jinan Central Hospital, Ji'nan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zigong Fourth People's Hospital, Zigong, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Luhe Hospital Capital Medical University, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Chongqing University Three Gorges Hospital, Chongqing
  - Tongji Hospital Affiliated to Tongji University, Shanghai
  - Shanghai East Hospital, Shanghai
  - Nankai Hospital of Tianjin City, Tianjin